CLINICAL TRIAL: NCT02100319
Title: Azilva Tablets Special Drug Use Surveillance "Hypertension Complicated by Diabetes "
Brief Title: Azilsaltan Tablets (Azilva Tablets) Special Drug Use Surveillance "Hypertension Complicated by Diabetes "
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 279-012; JapicCTI-142466 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-03-06; First posted 2014-03-31 (Estimated); Results first posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2018-12

CONDITIONS: Hypertension
Keywords: Pharmacological therapy
MeSH Terms: conditions — Hypertension | interventions — azilsartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Azilsartan at a dose of 20 to 40 mg, orally, once daily: Azilsartan tablets
  Interventions: Drug: Azilsartan

INTERVENTIONS:
Drug: Azilsartan — Azilsartan tablets
  Other Names: Azilva Tablets

SUMMARY:
The purpose of this study is to evaluate the efficacy of azilsartan tablets (Azilva Tablets) in patients with hypertension complicated by diabetes mellitus whose blood pressure cannot be sufficiently reduced by monotherapy with angiotensin II receptor blockers (ARBs) other than azilsartan, in routine clinical practice

DETAILED DESCRIPTION:
This study was designed to evaluate the efficacy of azilsartan tablets (Azilva Tablets) in patients with hypertension complicated by diabetes mellitus whose blood pressure cannot be sufficiently reduced by monotherapy with ARBs, other than azilsartan, in daily medical practice.

Patient enrollment will be started on April 1, 2014. The usual dosage for adults is 20 mg of azilsartan administered orally once daily. The dose can be adjusted according to the participant's age and condition. The maximum daily dose is 40 mg.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypertension who meet all the following criteria will be enrolled:

  1. Patients who has complications of diabetes mellitus
  2. Patients who is on monotherapy with ARBs (other than azilsartan) as antihypertensive treatment (Patients who have continued monotherapy with the same ARB product for at least 8 weeks at the time of Step-1* of participant enrollment and will continue such treatment until the first administration of Azilsartan Tablets)
  3. Patients who has a systolic blood pressure of ≥ 130 millimeter of mercury (mmHg) and/or diastolic blood pressure of 80 ≥ mmHg at the examination performed at the medical institution
  4. Patients who is an outpatient
  5. Patient who keeps a regular lifestyle and whose usual waking time is between 4 a.m. and 9:30 a.m.

     *For this surveillance, participant enrollment will be performed in two divided steps: Step-1 (at hospital visit before prescription of Azilsartan Tablets) and Step-2 (at the time of prescription of Azilsartan Tablets).

     Exclusion Criteria:
* Patients with contraindications to azilsartan

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hypertension
Sampling Method: Probability Sample
Enrollment: 387 (Actual)
Dates: Start 2014-03-03 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- Japan (2):
  - Osaka
  - Tokyo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 146 investigative sites in Japan, from 03 March 2014 to 29 February 2016.
Pre-assignment Details: Participants with a historical diagnosis of both hypertension and type 2 diabetes mellitus were enrolled. Participants received interventions as part of routine medical care.
Groups:
- Azilsartan 20 to 40 mg: Azilsartan 20 mg - 40 mg, tablet, orally, once daily for up to 24 weeks in participants based upon the disease severity. Participants received interventions as part of routine medical care.
Period: Overall Study
Arm/Group | Azilsartan 20 to 40 mg
Started | 387
Completed | 371
Not Completed | 16
Not completed — Case Report Forms Uncollected | 11
Not completed — Protocol Deviation | 5

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: The safety analysis set was defined as all participants who completed the study.
Arm/Group | Azilsartan 20 to 40 mg
Number analyzed (Participants) | 371
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.8 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150
  Male | 221
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Japan | 371
Type of Diabetes Mellitus [Count of Participants; unit: Participants]
  Type 1 Diabetes Mellitus | 2
  Type 2 Diabetes Mellitus | 369
Predisposition to Hypersensitivity [Count of Participants; unit: Participants] — The baseline characteristic was analyzed in participants who had a liability or tendency to suffer from hypersensitivity.
  Participants
    Had No Predisposition to Hypersensitivity | 345
    Had Predisposition to Hypersensitivity | 11
    Unknown | 15
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study excluding type 2 diabetes mellitus. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had No Presence of Medical Complications | 77
    Had Presence of Medical Complications | 294
Estimated Glomerular Filtration Rate (eGFR) [Count of Participants; unit: Participants] — Here "mL" is milliliter, "min" is minute, and "m" is meter. Population: The number analyzed is the number of participants with data available for analysis.
  Participants
    number analyzed (Participants) | 277
    >= 15 mL/min/1.73m^2 and < 30 mL/min/1.73m^2 | 4
    >= 30 mL/min/1.73m^2 and < 45 mL/min/1.73m^2 | 24
    >= 45 mL/min/1.73m^2 and < 60 mL/min/1.73m^2 | 57
    >= 60 mL/min/1.73m^2 and < 90 mL/min/1.73m^2 | 145
    >= 90 mL/min/1.73m^2 | 47
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  kg/m^2
    number analyzed (Participants) | 306
    (all) | 25.91 (4.667)
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 173
  Current Smoker | 48
  Ex-Smoker | 94
  Unknown | 56
Drinking Habits [Count of Participants; unit: Participants] — Participants who answered Yes or No for a question "Drink Alcohol Almost Every Day?" were reported
  Participants
    Yes | 73
    No | 241
    Unknown | 57
Pre-treatment ARB before Study Start [Count of Participants; unit: Participants] — ARB = Angiotensin II Receptor Blocker. Reported data was treatment drug of ARB before observational duration.
  Participants
    Losartan | 32
    Candesartan | 88
    Valsartan | 58
    Telmisartan | 89
    Olmesartan | 66
    Irbesartan | 38

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline in Blood Pressure on Final Assessment Point (up to Week 24) Measured at the Medical Institution
Description: Reported data were changes from baseline in blood pressure (systolic blood pressure [SBP] and diastolic blood pressure [DBP]) measured at the medical institution.
Time Frame: From baseline up to final assessment point (up to Week 24)
Population: Efficacy assessment population; The efficacy assessment population was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points available.
  The analyzed numbers were participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Millimeter of Mercury (mmHg)
Arm/Group | Azilsartan 20 to 40 mg
Number analyzed (Participants) | 371
Millimeter of Mercury (mmHg)
  Systolic Blood Pressure (SBP): number analyzed (Participants) | 355
  Systolic Blood Pressure (SBP) | -10.5 (18.40)
  Diastolic Blood Pressure (DBP): number analyzed (Participants) | 355
  Diastolic Blood Pressure (DBP) | -5.1 (11.57)

2. Primary Outcome: Changes From Baseline in Home Blood Pressure on Final Assessment Point (up to Week 24)
Description: Reported data were changes from baseline in blood pressure (SBP and DBP) measured at home right after waking up and at bedtime.
Time Frame: From baseline up to final assessment point (up to Week 24)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan 20 to 40 mg
Number analyzed (Participants) | 371
mmHg
  SBP Right after Waking-up: number analyzed (Participants) | 246
  SBP Right after Waking-up | -7.9 (14.86)
  DBP Right after Waking-up: number analyzed (Participants) | 246
  DBP Right after Waking-up | -4.1 (8.07)
  SBP at Bedtime: number analyzed (Participants) | 138
  SBP at Bedtime | -7.1 (13.82)
  DBP at Bedtime: number analyzed (Participants) | 138
  DBP at Bedtime | -4.3 (7.76)

3. Secondary Outcome: Changes From Baseline in Pulse Rate on Final Assessment Point (up to Week 24) at the Medical Institution
Description: Reported data were changes from baseline in pulse rate measured at the medical institution.
Time Frame: From baseline up to final assessment point (up to Week 24)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Beat per Minutes (bpm)
Arm/Group | Azilsartan 20 to 40 mg
Number analyzed (Participants) | 371
Beat per Minutes (bpm) | -1.3 (10.22)

4. Secondary Outcome: Changes From Baseline in Hemoglobin A1c (HbA1c) on Final Assessment Point (up to Week 24) at the Medical Institution
Description: Reported data were changes from baseline in HbA1c (National glycohemoglobin standardization program [NGSP] value) measured at the Medical Institution.
Time Frame: From baseline up to final assessment point (up to Week 24)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Azilsartan 20 to 40 mg
Number analyzed (Participants) | 371
Percent | 6.72 (0.792)

5. Secondary Outcome: Changes From Baseline in Creatinine-adjusted Urinary Albumin Level on Final Assessment Point (up to Week 24) at the Medical Institution
Description: Reported data were changes from baseline in creatinine-adjusted urinary albumin level (that is calculated from urinary albumin level divided by creatinine level) measured at the medical institution. Here "mg/gCr" is Milligrams per Gram of Creatinine.
Time Frame: From baseline up to final assessment point (up to Week 24)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/gCr
Arm/Group | Azilsartan 20 to 40 mg
Number analyzed (Participants) | 371
mg/gCr | -44.344 (413.9519)

6. Secondary Outcome: Percentage of Participants Who Had One or More Adverse Events
Time Frame: Up to Week 24
Population: Safety Analysis Set; The safety analysis set was defined as all participants who completed the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | Azilsartan 20 to 40 mg
Number analyzed (Participants) | 371
Percentage of Participants | 6.47

ADVERSE EVENTS:
Time Frame: Up to Week 24
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Azilsartan 20 to 40 mg
All-Cause Mortality (participants affected / at risk) | 2/371
Serious Adverse Events (participants affected / at risk) | 5/371
Other Adverse Events (participants affected / at risk) | 20/371
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan 20 to 40 mg (N=371)
Sepsis (Infections and infestations) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Sudden death (General disorders) | 1 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan 20 to 40 mg (N=371)
Diabetes mellitus (Metabolism and nutrition disorders) | 7
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1
Dizziness postural (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Feeling abnormal (General disorders) | 1
Oedema peripheral (General disorders) | 1
Blood pressure increased (Investigations) | 2
Blood glucose increased (Investigations) | 1
Glycosylated haemoglobin increased (Investigations) | 3
Blood creatinine increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.